CLINICAL TRIAL: NCT03482674
Title: DIMINI - Activating of Health Literacy in Persons With an Increased Risk of Type 2 Diabetes Mellitus by Coaching at General Practitioners
Brief Title: DIMINI - Diabetes Mellitus? - Not me!
Acronym: Dimini
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dimini Konsortium (Other)
Collaborators: Deutsche Diabetes Gesellschaft (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 01NVF17012
Record Dates: First submitted 2018-03-06; First posted 2018-03-29 (Actual); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Health Behavior; Health Knowledge, Attitudes, Practice; Literacy; Diabetes Mellitus, Type 2; Diabetes
Keywords: Health literacy; Innovation Fund; lifestyle intervention; risk screening; type 2 diabetes mellitus; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Health Behavior; Behavior; Literacy; Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): The control group will receive standard care as provided by the German statutory health insurance.
- Intervention group (Experimental): The intervention group receives the DIMINI lifestyle intervention for a period of three months.
  Interventions: Behavioral: DIMINI lifestyle intervention

INTERVENTIONS:
Behavioral: DIMINI lifestyle intervention — DIMINI lifestyle intervention consists of the DIMINI-kit which contains health information, a list of food recommendations with additional information on calories, serving size and weight (traffic light rating system), a nutrition and an exercise diary. Participants in the intervention group can choose between a paper-based version or an app-based version of the DIMINI-kit. In addition, the kit includes an elastic exercise band with exercise poster, a measuring tape for self-control of the waist size and a pedometer.
  Arms: Intervention group

SUMMARY:
The increasing prevalence of type 2 diabetes mellitus is a worldwide problem. In preventing risk factors and unhealthy lifestyle through improved health literacy, chances are seen to delay or even avoid type 2 diabetes mellitus. The aim of the DIMINI-project is to prevent type 2 diabetes mellitus and to strengthen the health literacy of people at increased risk of developing it. For this purpose, people at increased risk are first identified by using the standardized screening tool Finnish Diabetes Risk Score (FINDRISC) adapted for Germany. Identified risk persons then receive a needs-based, modular lifestyle intervention including nutrition tips and physical exercises either paper- or app-based.

DETAILED DESCRIPTION:
DIMINI, a randomised controlled trial, will assess whether the implementation of a lifestyle intervention for people at increased risk of developing type 2 diabetes mellitus will result in an improvement in body weight (primary outcome) and participants health literacy (secondary outcome) or not. A three-month intervention in the intervention group is followed by a one-year follow-up. The control group receives standard care as provided by the German statutory health insurance for three months and a one-year follow-up as well.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* resident in Hesse or Schleswig-Holstein
* statutory health insurance in one out of five participating health insurances
* overweight/obesity
* low physical activity
* known family disposition for type 2 diabetes mellitus
* history of increased glucose levels
* FINDRISC results with scores ≥ 12

Exclusion Criteria:

* age < 18 years
* resident outside Hesse or Schleswig-Holstein
* statutory or private health insurance with other than the participating health insurances
* clinically manifested diabetes mellitus
* malnutrition
* psychiatric disorders
* pregnancy
* FINDRISC results with scores <12
* participation in other clinical trials

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 530 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Body weight reduction | 15 Months
  Survey of weight general practitioners level

SECONDARY OUTCOMES:
Health literacy (European Health Literacy Survey Questionnaire) | 15 Months
  Summed scale:
  * Maximum: 16 (best health literacy)
  * Minimum: 0 (worst health literacy)
  * ≥ 13 = sufficient health literacy
  * 9-12 = problematic health literacy
  * ≤ 8 = inadequate health literacy Higher values represent a better outcome
Eating behaviour (German questionnaire on eating behaviour) | 15 Months
  Three summed subscales:
  Scale 1) cognitive control of eating behavior, restrained eating
  * Minimum score: 0 = no cognitive control
  * Maximum score: 21 = extreme cognitive control Scale 2) disturbance of eating behavior
  * Minimum score: 0 = no disturbance
  * Maximum score: 16 = extreme disturbance Scale 3) experienced feelings of hunger
  * Minimum score: 0 = no disturbing sensations of hunger
  * Maximum score: 14 = very strong disturbing sensations of hunger For each item it is determined individually, which response option is considered to get a value of 1 or a value of 0 (e.g. Scale 1 Item 12: "true" = 1, "not true" = 0, Item 18 "true" = 0, "not true" = 1)
Physical activity (International Physical Activity Questionnaire) | 15 Months
  Questionnaire designed for population surveillance of physical activity among adults including
  Total Score:
  * Maximum Score: 960 minutes
  * Minimum Score: 10 minutes
  Categorical Score:
  Category 1 - Low:
  • Individuals who not meet criteria for Categories 2 or 3
  Category 2 - Moderate:
  * 3 or more days of vigorous-intensity activity of at least 20 minutes per day
  * 5 or more days of moderate-intensity activity and/or walking of at least 30 minutes per day
  * 5 or more days of any combination of walking, moderate-intensity or vigorous intensity activities achieving a minimum total physical activity of at least 600 minutes/week.
  Category 3 High
  * vigorous-intensity activity on at least 3 days achieving a minimum total physical activity of at least 1500 minutes/week
  * 7 or more days of any combination of walking, moderate-intensity or vigorous-intensity activities achieving a minimum total physical activity of at least 3000 minutes/week.
Quality of life | 15 Months
  Short Form 12

CONTACTS AND LOCATIONS:
Overall Officials: Carsten Petersen, Dr., Principal Investigator — docevent GmbH
Locations (1):
- docevent GmbH, Schleswig, Schleswig-Holstein, Germany

REFERENCES:
- [Derived] Puschner F, Wetzel S, Urbanski-Rini D, Bertram N, Schliffke M, Gohl M, Petersen C; Dimini Consortium. The association between the risk of developing type 2 diabetes mellitus and health-related quality of life: baseline results from the Dimini lifestyle intervention. Qual Life Res. 2021 Dec;30(12):3523-3533. doi: 10.1007/s11136-021-02878-2. Epub 2021 May 19. PMID 34008163